CLINICAL TRIAL: NCT03211260
Title: Effects of Proprioceptive Focal Stimulation (EQUISTASI) on Freezing of Gait in Parkinson's Disease: a Open, Single-arm Trial
Brief Title: Effects of Proprioceptive Focal Stimulation (EQUISTASI) on Freezing of Gait in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Iterim analysis did not detect a clinically meaningful change in the primary endpoint
Sponsor: ASST Gaetano Pini-CTO (Other)
Collaborators: Grisons Foundation for Parkinson's Disease (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gianni Pezzoli, Principal Investigator, ASST Gaetano Pini-CTO
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 319_2017bis
Record Dates: First submitted 2017-07-02; First posted 2017-07-07 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Freezing of Gait; Parkinson Disease
Keywords: Parkinson Disease; Freezing of gait; Equistasi
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EQUISTASI (Experimental): Equistasi is a nanotechnology for proprioceptive focal stimulation. Every patient will receive four patches to be placed on both legs for 4 weeks.
  Interventions: Device: EQUISTASI

INTERVENTIONS:
Device: EQUISTASI — Equistasi is a nanotechnology for proprioceptive focal stimulation. Every patient will receive four patches to be placed on both legs for 4 weeks.

SUMMARY:
Freezing of gait (FOG) is a common disabling condition in Parkinson's disease (PD), causes falls, and impairs quality of life. Therapeutic options for this symptom are limited and of limited efficacy. Besides, the pathophysiology has been not clarified yet. Proprioceptive sensitivity is likely to play a role and recent studies have reported that high-frequency microfocal vibratory stimulation exert a modulatory effect of proprioceptive reflex circuits and could be considered a valuable treatment strategy. However, evidence is not available. The present study was designed to collect preliminary evidence of efficacy of a vibrotactile device (Equistasi) for the treatment of FOG.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's Disease
* Stable drug therapy response without any change in the 3 months before the study.
* written informed consent

Exclusion Criteria:

* Hoehn-Yahr stage ≥ 4
* Cognitive decline (Mini Mental State Examination <26)
* Systemic illness involving the nervous system
* Diabetes
* Presence of cardiac pacemaker
* Presence of deep brain stimulation
* Presence of severe dysautonomia with marked hypotension
* History or active neoplasia
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Freezing of gait questionnaire severity | 4 weeks
  Change in freezing of gait questionnaire score

SECONDARY OUTCOMES:
Gait and Falls Questionnaire (GFQ) score | 4 weeks
  Change in the GFQ score
39-item Parkinson's Disease Questionnaire | 4 weeks
  Change in quality of life measured using the 39-item Parkinson's Disease Questionnaire
Falls | 4 weeks
  Number of falls recorded during the intervention period
Treatment continuation | 4 weeks
  Likelihood that patients would continue taking the trial treatment as assessed by a self-rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Pezzoli, MD, Principal Investigator — Centro Parkinson, ASST Gaetano Pini-CTO di Milano
Locations (1):
- Centro Parkinson, ASST Gaetano Pini-CTO, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided